CLINICAL TRIAL: NCT02866539
Title: A Polyherbal for Control of Blood Sugar in Subjects With Impaired Glucose Tolerance and/or Early Type 2 Diabetes. A Randomized Placebo Controlled Study of a Polyherbal (Whole Herb Formulation)
Brief Title: Effect of Polyherbal Compound for Control of Blood Sugar in Impaired Glucose Tolerance and Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Composite Interceptive Med Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OI - 001 - 2016
Record Dates: First submitted 2016-08-04; First posted 2016-08-15 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polyherbal capsule (Active Comparator): Polyherbal capsule contains leaves of 3 herbs namely C. indica, B. spectabilis and C. rosea.
  Interventions: Drug: Polyherbal capsule coccinia, bougainvillea, catharanthus
- Placebo (Placebo Comparator): Placebo will contain an inert substance
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Polyherbal capsule coccinia, bougainvillea, catharanthus — A unique combination of 3 herbs that lower blood sugars
  Other Names: Sugar Balance (SB)
  Arms: Polyherbal capsule
Drug: Placebo — Similar looking inactive powder
  Arms: Placebo

SUMMARY:
The aim of the study is to control blood sugar with Sugar Balance capsules which is the leaves of three herbs: ivy ground (Coccinia indica)-200mg, bougainvillia (Bougainvillea spectabilis)-30mg, Madagascar periwinkle (Catharanthus rosea)-20mg.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and non-pregnant females aged ≥30 years having a diagnosis of pre-diabetes (impaired fasting glucose or impaired glucose tolerance) and a diabetes and a meeting one of the following criteria

  1. Fasting Plasma Glucose ≥100 mg/dL, fasting is defined as no caloric intake for at least 8 h, OR
  2. 2-h Post load Glucose ≥140 mg/dL during an Oral Glucose Tolerance Test (OGTT). The test should be performed as described by the World Health Organisation(WHO), using a glucose load containing the equivalent of 75 g anhydrous glucose dissolved in water. OR
  3. Glycosylated haemoglobin (A1C) ≥5.7%. The test should be performed in a laboratory using a method that is National Accreditation Board for Testing and Calibration Laboratories certified and standardized. OR
  4. In a patient with classic symptoms of hyperglycaemia or hyperglycaemic crisis, a random plasma glucose ≥200 mg/dL in the last 12 months.

Exclusion Criteria:

* Any one of the following

  1. History of diabetes onset >12 months from date of randomization and/or on any oral hypoglycemic agents (other than metformin)
  2. Any history suggestive of micro vascular or macro vascular disease
  3. Women in childbearing age unable to practice any form of contraception
  4. Impaired renal function; estimated glomerular filtration rate(eGFR) <60mls/min/1.73m2.
  5. Known history of any chronic illness taking regular pharmacological agents.
  6. Blood pressure fluctuations exceeding 10 mmHg on 2 subsequent clinic visits or known history of hypotension or bradycardia in last 6 months or taking 2 or more antihypertensive medications regularly in the last 6 weeks
  7. Current or former employees of organic India
  8. Participating in another clinical trial with an active intervention or drug or device with last dose taken within 60 days.
  9. Refusing consent or physician uncomfortable with patient compliance to treatments or follow up.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2016-12; Primary Completion 2017-12-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Number of diabetes subjects achieving glycemic control | 6 months
  a 0.5% reduction in baseline A1c and/or fasting plasma glucose below 125 mg/dl or 2 hour postprandial glucose <180 mg/dl
Number of pre-diabetes achieving euglycemic status | 6 months
  measured as A1c < 5.7% and/or fasting plasma glucose <100mg/dl/

CONTACTS AND LOCATIONS:
Overall Officials: Alben Sigamani, MD, Principal Investigator — Narayana Hrudayalaya Hospital
Locations (1):
- Narayana Hrudayalaya Limited, Mazumdar Shaw multispecialty Hospital, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided